CLINICAL TRIAL: NCT02699762
Title: Randomised Controlled Trial to Evaluate the Effect of a Self-rehabilitation Program in Addition to Usual Treatment for Spasticity on Upper Limb Function in Stroke
Brief Title: Upper Limb Botulinum Toxin Injection Combined With Self Rehabilitation
Acronym: Armautotox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2015-A01677-42
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-01

CONDITIONS: Self Rehabilitation Combined With BTI on Upper Limb
Keywords: self rehabilitation; stroke; botulinum toxin injection; arm functions
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): self rehabilitation of upper limb in experimental group + BTI + usual physiotherapy
  Interventions: Other: self rehabilitation of upper limb in experimental group
- control group (No Intervention): BTI + usual physiotherapy

INTERVENTIONS:
Other: self rehabilitation of upper limb in experimental group — The patients in the self-rehabilitation group will be taught the self-rehabilitation program by a physiotherapist who is not involved in the patient follow-up. They will receive a log book which will be used to evaluate compliance and tolerance to the program. They will be instructed to carry out the exercises 7 days per week for the whole duration of the study and to record which exercises they carried out and for how long, after each exercise session.
  Arms: experimental group

SUMMARY:
To show that the addition of a self-rehabilitation program to standard treatment, involving repeated BTI and usual physiotherapy, improves impairment and activity limitation of the paretic upper limb more than the control treatment (BTI + usual physiotherapy), in a randomised controlled study of patients with spastic hemiparesis following stroke.

DETAILED DESCRIPTION:
Following stroke, 30% of patients are left with a "hemiplegic" upper limb meaning that they are unable to carry out any movements with the limb and are thus partially or totally dependent for all activities of daily living (dressing, washing, feeding etc). Another 40% have some proximal recovery. These patients are able to carry out some movement of the shoulder and sometimes the elbow. They can use the limb for some activities of daily living such as carrying a bag or stabilising paper while writing. The last 30% recover a certain degree of prehension, however their motor control is altered and they have impairments of both the reaching and grasping phases.

Treatment for chronic stroke symptoms (more than 6 months post-onset) including impairments and activity limitations is mostly based on physiotherapy and botulinum toxin injections (BTI).

Physiotherapy : This treatment has been shown to be effective, and is essential to reduce impairments and improve function in patients with hemiparesis following stroke (Robertson et al, 2008 ; Bourgeais et al, 2010). Different methods exist, and comparative studies of the most common ones have shown a similar effectiveness (Adal et al, 2006 ; Flansbjer et al, 2008 ; Brazzelli et al, 2011, Durstine et al 2009). No conventional treatment has been shown to be more effective than another. However, it has been demonstrated that the intensity and specificity of rehabilitation techniques are positively correlated with motor recovery (Gordon et al, 2004).

Intensity of rehabilitation: In 2006, a meta-analysis of 21 studies on the effect of muscle strengthening post stroke showed that it improved active function and activities of daily living (measured on different scales) following acute and chronic stroke (Ada et al, 2006). Currently, a meta-analysis by Brazzelli et al. (2011) contains the largest collection of data, with 32 studies and a total of 1414 participants. The studies included were on the subject of cardiovascular training, muscle strengthening and mixed training (cardiovascular+strength). The main outcome measures were the incidence of mortality and the degree of dependence and disability. The results showed improvements following cardiovascular training and mixed training. Strength training alone did not significantly improve mobility. These results lead the American College of Sport and Medicine to recommend endurance and strength training coupled with stretching for stroke patients.

Task-oriented training : Carr et Shepherd (1998) were the first to promote task oriented training. More recently, Van de port et al, (2009-2012) evaluated 250 patients following 12 weeks of task-oriented circuit training (126 patients) or conventional physiotherapy (124 patients). All the patients were at least 6 months post stroke. The training consisted of 6-minute work stations with 8 different exercises, such as rising from a chair to reach different targets, picking up objects from the floor while walking, kicking a ball, crossing obstacles, ascending and descending stairs etc. Greater improvements occurred in the task-oriented group for the six-minute walk test and the Stair test (time to ascend and descend a flight of 10 stairs. Another meta-analysis (including 307 participants) demonstrated that task-oriented training improves distance walked, gait speed and the Timed Up and Go test (rising from a chair, walking 3 metres, turning and returning to sit) (Wevers et al, 2009). These results show that training should involve practice of the specific function to be improved.

Botulinum toxin injections : Botulinum toxin is a neurotoxin produced by the clostridium botulinum bacteria. Seven different serotypes exist but only the A and B serotypes are used in clinical practice. Botulinum toxin blocks the presynaptic release of neurotransmitter at the neuromuscular junction. Focal transitory paralysis thus occurs in the injected muscle. Its action lasts on average 3 months in striated skeletal muscle. The effect of BTI in the upper limb depends on the parameters studied. A meta-analysis carried out by Foley et al, 2013 showed a relatively large effect size for the reduction of impairment and the improvement of passive function. However, there was only a small effect size for the improvement of functions such as prehension. This confirms the results of a previous study (Sheean et al, 2010) which showed that the effect of BTI in the upper limb was only significant for the reduction of impairment or the improvement of passive function, but not active function.

These results were further confirmed in a study which used goal attainment scaling as an outcome measure (Turner Stokes et al, 2010). Following BTI in the upper limb of hemiparetic patients, there was a significant improvement in the goal attainment scaling score which was, moreover, strongly correlated with the reduction in spasticity evaluated with the Ashworth scale (most widely used scale for the evaluation of spasticity). The results also showed that the goal was more often attained when it involved the improvement of a passive function than an active function. The only study to have shown an improvement in prehension following BTI involved combined treatment with constraint induced therapy (Sun et al, 2010).

Self-rehabilitation Two recent studies have shown that rehabilitation coupled with BTI could have a significant effect on activity limitation: A pilot randomised controlled trial of 35 patients with spastic hemiparesis by Roche et al (2014) showed that a 30-minute, daily self-rehabilitation program coupled with a single session of BTI in the lower limb significantly improved several gait-related activities. The self-rehabilitation program was developed to combine different types of exercises including: i) strengthening of the hip flexors and extensors and the triceps sural; ii) stretching of the rectus femoris, hamstrings and triceps sural and iii) task-oriented gait-related exercises including obstacle crossing and slaloming. They showed significantly greater improvements in the experimental group than the control group for maximal gait speed in the 10-metre walk test, distance walked in the 6-minute walk test and the time to ascend and descend a flight of stairs. Sun et al (2010) carried out a randomised controlled trial which included 32 patients with stroke. They showed that constraint-induced therapy in the paretic upper limb coupled with BTI significantly improved prehension and reduced spasticity in the finger and wrist flexors more than BTI coupled with standard therapy.

In summary Together, these results indicate that the addition of a self-rehabilitation program to botulinum toxin injections is the most pertinent method to optimise the effects of BTI and usual therapy. However, no study has yet evaluated the effects of the addition of a self-rehabilitation program to treatment by BTI and usual therapy.

Moreover, this corresponds to a public health issue which is to provide a greater intensity of rehabilitation within the constraints of the health system, including lack of funding and lack of physiotherapists trained in this type of specialised rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged from 18 to 75 years inclusive.
* Women at least 24 months post menopause, or having undergone surgical sterilisation or using an effective method of contraception (oral or injected contraception or patches or a double-barrier intrauterine device).
* Signing of the informed consent form indicating that the subject has understood the aim of the study as well as the procedures involved and that he/she accepts to participate and to comply with the demands and restrictions inherent to the study
* Affiliation to the French social security regime or a similar regime.
* Single stroke more than 6 months previously
* Capable of understanding instructions and to participate in the definition of a therapeutic goal
* Voluntary movement of the shoulder and elbow
* Able to participate in a self-rehabilitation program
* Having previously undergone BTI. The last injection must be at least 4 months prior to inclusion.

Exclusion Criteria:

* Subjects who are unlikely to adhere to the study and/or poor adherence anticipated by the investigator
* Patient with no medical insurance
* Pregnant woman
* Uncontrolled progressive pathology
* Comprehension deficit (Boston Diagnostic Aphasia Examination(BDAE) <3)
* Osteoarticular lesion which contraindicates part of the rehabilitation involved in the study
* Patients with other interventions planned prior to the end of the study period (orthosis, surgery etc.)
* Surgery to the paretic limb treated in the study less than 6 months previously
* Contra-indications to botulinum toxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
wolf-motor functional test (WMFT) | 1h
  functional hemiplegic's arm evaluation

SECONDARY OUTCOMES:
modified Ashworth scale | 15 minutes
  spasticity evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD PhD, Principal Investigator — Raymond Poincare HOSPITAL
Locations (1):
- Raymond Poincare Hospital, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maulet T, Pouplin S, Bensmail D, Zory R, Roche N, Bonnyaud C. Self-rehabilitation combined with botulinum toxin to improve arm function in people with chronic stroke. A randomized controlled trial. Ann Phys Rehabil Med. 2021 Jul;64(4):101450. doi: 10.1016/j.rehab.2020.10.004. Epub 2020 Dec 17. PMID 33152520